CLINICAL TRIAL: NCT04344340
Title: The Association Between MIH and HSPM
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yassmin Mohamed Abdelrahman, principle invistigator, Cairo University
Other Study IDs: MIH and HSPM
Record Dates: First submitted 2020-03-06; First posted 2020-04-14 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Hypomineralization of Enamel; Hypomineralization Molar Incisor
Keywords: HSPM & MIH
MeSH Terms: conditions — Dental Enamel Hypomineralization; Molar Hypomineralization | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: clinical examination — clinical examination

SUMMARY:
Aim of the Study Evaluate association between HSPM and MIH in Egyptian children. Record the prevalence of HSPM and MIH in Egyptian children

DETAILED DESCRIPTION:
Statement of the Problem:

Molar Incisor Hypomineralization (MIH) is defined as developmental qualitative defect of systemic origin, which affects one to four of first permanent molars and frequently associated with permanent incisors . The prevalence of MIH worldwide was reported from 2.4% to40.2% and clinical measures of MIH based on scientific criteria was established based on the European Academy of Pediatric Dentistry criteria to allow comparison between the findings of different studies .

The most commonly reported clinical problems for patients with MIH are hypersensitivity of teeth to various thermal and mechanical stimuli result in improper tooth brushing, plaque accumulation and rapid caries progression. Severely affected enamel shows post eruptive breakdown and such teeth require extensive treatment, ranging from prevention to restorations and extractions. MIH patients also have increased risk of developing dental fear and anxiety as well as behavior management problems added to the difficulty to achieve effective local anaesthesia which are related to chronic pulp inflammation from dentin exposure due to excessive enamel breakdown.

Rational As developmental of Second Primary Molar start at the same time as the development of the first permanent molars and incisor but the maturation of permanent teeth occur more slow. So when a systemic disturbance occur it affect second primary molar as well as first permanent molar and incisors.

Few studies test the association between hypomineralized second primary molar (HSPM) and MIH. While no study available on Egyptian children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 8 to 9 years.
* Both genders.
* No systemic health problems

Exclusion Criteria:

* Children with extracted primary second molars and permanent incisors and molars.
* Children with history of dental trauma.
* Children with orthodontic bands or dental appliances

Ages: 8 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: Healthy children aged from 8 to 9 years attending outpatient clinic in Pediatric Dentistry Department, Faculty of Dentistry, Cairo University will be included in this study according to eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of hypomineralized second primary molars. | 1 year
  The percentage of children who has enamel defect on their second primary molars in the study

SECONDARY OUTCOMES:
the prevalence of Molar Incisor Hypomineralization | 1 year
  The percentage of children who has enamel defect on their permenant molars and Incisors at this study

CONTACTS AND LOCATIONS:
Overall Officials: Rania A Taha, Professor, Study Director — Cairo U
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Broadbent JM, Thomson WM, Williams SM. Does caries in primary teeth predict enamel defects in permanent teeth? A longitudinal study. J Dent Res. 2005 Mar;84(3):260-4. doi: 10.1177/154405910508400310. PMID 15723867
- [Background] Elfrink ME, ten Cate JM, Jaddoe VW, Hofman A, Moll HA, Veerkamp JS. Deciduous molar hypomineralization and molar incisor hypomineralization. J Dent Res. 2012 Jun;91(6):551-5. doi: 10.1177/0022034512440450. Epub 2012 Feb 27. PMID 22370445
- [Background] Elfrink ME, Schuller AA, Weerheijm KL, Veerkamp JS. Hypomineralized second primary molars: prevalence data in Dutch 5-year-olds. Caries Res. 2008;42(4):282-5. doi: 10.1159/000135674. Epub 2008 Jun 4. PMID 18523388
- [Background] Elfrink ME, Ghanim A, Manton DJ, Weerheijm KL. Standardised studies on Molar Incisor Hypomineralisation (MIH) and Hypomineralised Second Primary Molars (HSPM): a need. Eur Arch Paediatr Dent. 2015 Jun;16(3):247-55. doi: 10.1007/s40368-015-0179-7. Epub 2015 Apr 18. PMID 25894247
- [Background] Garot E, Denis A, Delbos Y, Manton D, Silva M, Rouas P. Are hypomineralised lesions on second primary molars (HSPM) a predictive sign of molar incisor hypomineralisation (MIH)? A systematic review and a meta-analysis. J Dent. 2018 May;72:8-13. doi: 10.1016/j.jdent.2018.03.005. Epub 2018 Mar 14. PMID 29550493
- [Background] Ghanim A, Manton D, Marino R, Morgan M, Bailey D. Prevalence of demarcated hypomineralisation defects in second primary molars in Iraqi children. Int J Paediatr Dent. 2013 Jan;23(1):48-55. doi: 10.1111/j.1365-263X.2012.01223.x. Epub 2012 Jan 25. PMID 22276809
- [Background] Ghanim A, Elfrink M, Weerheijm K, Marino R, Manton D. A practical method for use in epidemiological studies on enamel hypomineralisation. Eur Arch Paediatr Dent. 2015 Jun;16(3):235-46. doi: 10.1007/s40368-015-0178-8. Epub 2015 Apr 28. PMID 25916282
- [Background] Ghanim A, Silva MJ, Elfrink MEC, Lygidakis NA, Marino RJ, Weerheijm KL, Manton DJ. Molar incisor hypomineralisation (MIH) training manual for clinical field surveys and practice. Eur Arch Paediatr Dent. 2017 Aug;18(4):225-242. doi: 10.1007/s40368-017-0293-9. Epub 2017 Jul 18. PMID 28721667
- [Background] Leppaniemi A, Lukinmaa PL, Alaluusua S. Nonfluoride hypomineralizations in the permanent first molars and their impact on the treatment need. Caries Res. 2001 Jan-Feb;35(1):36-40. doi: 10.1159/000047428. PMID 11125194
- [Background] Lygidakis NA, Dimou G, Marinou D. Molar-incisor-hypomineralisation (MIH). A retrospective clinical study in Greek children. II. Possible medical aetiological factors. Eur Arch Paediatr Dent. 2008 Dec;9(4):207-17. doi: 10.1007/BF03262637. PMID 19054474
- [Background] Negre-Barber A, Montiel-Company JM, Boronat-Catala M, Catala-Pizarro M, Almerich-Silla JM. Hypomineralized Second Primary Molars as Predictor of Molar Incisor Hypomineralization. Sci Rep. 2016 Aug 25;6:31929. doi: 10.1038/srep31929. PMID 27558479
- [Background] Weerheijm KL, Jalevik B, Alaluusua S. Molar-incisor hypomineralisation. Caries Res. 2001 Sep-Oct;35(5):390-1. doi: 10.1159/000047479. No abstract available. PMID 11641576
- [Background] Weerheijm KL, Mejare I. Molar incisor hypomineralization: a questionnaire inventory of its occurrence in member countries of the European Academy of Paediatric Dentistry (EAPD). Int J Paediatr Dent. 2003 Nov;13(6):411-6. doi: 10.1046/j.1365-263x.2003.00498.x. PMID 14984047
- [Background] Butler PM. Comparison of the development of the second deciduous molar and first permanent molar in man. Arch Oral Biol. 1967 Nov;12(11):1245-60. doi: 10.1016/0003-9969(67)90126-4. No abstract available. PMID 5234231
- [Background] Whatling R, Fearne JM. Molar incisor hypomineralization: a study of aetiological factors in a group of UK children. Int J Paediatr Dent. 2008 May;18(3):155-62. doi: 10.1111/j.1365-263X.2007.00901.x. PMID 18384347
- [Background] Small BW, Murray JJ. Enamel opacities: prevalence, classifications and aetiological considerations. J Dent. 1978 Mar;6(1):33-42. doi: 10.1016/0300-5712(78)90004-0. No abstract available. PMID 275292